CLINICAL TRIAL: NCT00114400
Title: B-Vitamin Atherosclerosis Intervention Trial (BVAIT)
Brief Title: BVAIT: B-Vitamin Atherosclerosis Intervention Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Leiner Health Products (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG0024; R01AG017160 (NIH)
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2007-02

CONDITIONS: Atherosclerosis
Keywords: cardiovascular disease; CVD
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Folic Acid; Vitamin B 12; Vitamin B 6

INTERVENTIONS:
Drug: folic acid
Drug: vitamin B12
Drug: vitamin B6

SUMMARY:
The purpose of this study is to examine whether vitamin B supplementation will reduce the progression of early atherosclerosis in individuals over 40 years old and without clinical evidence of cardiovascular disease (CVD).

DETAILED DESCRIPTION:
The primary hypothesis to be tested is that daily vitamin B supplementation reduces progression of early atherosclerosis. Ultrasonography will be used to measure the rate of change in the thickness of the carotid artery and CT will be used to measure coronary and aortic calcium. The beneficial effects of vitamin B supplementation are expected to occur with or without a change in LDL-C levels.

A total of 506 men and women will be randomized to receive either 1) vitamin B supplementation consisting of folic acid 5mg, vitamin B12 0.4mg, and vitamin B6 50mg, or 2) a matching placebo. Participants will receive ultrasonography at baseline and every 6 months for 2.5 to 4.5 years, and CT scan at baseline and end of study (2.5 to 4.5 years).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (postmenopausal)
* 40 years or older
* Fasting plasma homocysteine 8.5 micromoles per liter (µmol/L) or greater

Exclusion Criteria:

* Any clinical signs or symptoms of cardiovascular disease (CVD)
* Diabetes mellitus or fasting serum glucose 140 mg/dL or greater
* Triglyceride (TG) levels 500mg/dL or greater
* Serum creatinine greater than 1.6 mg/dL
* Uncontrolled hypertension (systolic blood pressure 160 mmHg or greater and/or diastolic blood pressure 100 mmHg or greater)
* Thyroid disease (untreated)
* Life threatening disease with prognosis less than 5 years
* Alcohol intake greater than 5 drinks per day (1 drink = 1 1/2 oz distilled spirits, 4 oz wine, or 12 oz beer) or substance abuse (intravenous drug use, cocaine use)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 506
Dates: Start 2000-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
rate of change of distal common carotid artery (CCA) far wall intima-media thickness (IMT)

SECONDARY OUTCOMES:
change in coronary and abdominal aortic calcification
neurocognitive change

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, MD, Principal Investigator — University of Southern California, Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine
Locations (1):
- Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine, Los Angeles, California, United States

REFERENCES:
- [Derived] Lin F, Pa J, Karim R, Hodis HN, Han SD, Henderson VW, St John JA, Mack WJ. Subclinical carotid artery atherosclerosis and cognitive function in older adults. Alzheimers Res Ther. 2022 May 7;14(1):63. doi: 10.1186/s13195-022-00997-7. PMID 35526057
- [Derived] Hodis HN, Mack WJ, Dustin L, Mahrer PR, Azen SP, Detrano R, Selhub J, Alaupovic P, Liu CR, Liu CH, Hwang J, Wilcox AG, Selzer RH; BVAIT Research Group. High-dose B vitamin supplementation and progression of subclinical atherosclerosis: a randomized controlled trial. Stroke. 2009 Mar;40(3):730-6. doi: 10.1161/STROKEAHA.108.526798. Epub 2008 Dec 31. PMID 19118243